CLINICAL TRIAL: NCT03296527
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multicentre, Pan-Asian Trial Comparing the Efficacy and Safety of FE 999049 With Follitropin Alfa (GONAL-F) in Controlled Ovarian Stimulation in Women Undergoing Assisted Reproductive Technology Programme
Brief Title: Efficacy and Safety of FE 999049 in Controlled Ovarian Stimulation in Pan-Asian Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000145
Record Dates: First submitted 2017-09-14; First posted 2017-09-28 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2021-04

CONDITIONS: Controlled Ovarian Simulation
MeSH Terms: interventions — follitropin alfa; follitropin delta; FE 999049

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follitropin delta (Experimental): Recombinant follicle-stimulating hormone (rFSH). Follitropin delta for subcutaneous injection
  Interventions: Drug: Follitropin delta
- Gonal-F (Active Comparator): rFSH. Follitropin alfa for subcutaneous injection
  Interventions: Drug: Follitropin alfa

INTERVENTIONS:
Drug: Follitropin alfa — GONAL-F dose was fixed for the first 5 stimulation days.
  Other Names: GONAL-F
  Arms: Gonal-F
Drug: Follitropin delta — REKOVELLE (FE 999049) was fixed throughout the stimulation period.
  Other Names: FE 999049; REKOVELLE
  Arms: Follitropin delta

SUMMARY:
To demonstrate non-inferiority of FE 999049 compared with GONAL-F with respect to ongoing pregnancy rate in women undergoing controlled ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Documents signed prior to screening evaluations.
* In good physical and mental health in the judgement of the investigator.
* Asian pre-menopausal females between the ages of 20 and 40 years. The participants must be at least 20 years (including the 20th birthday) when they sign the informed consent and no more than 40 years (up to the day before the 41st birthday) at the time of randomization.
* Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II (defined by the revised American Society for Reproductive Medicine [ASRM] classification, 1996) or with partners diagnosed with male factor infertility, eligible for in vitro fertilisation (IVF) and/or intracytoplasmic sperm injection (ICSI) using fresh or frozen ejaculated sperm from male partner or sperm donor.
* Infertility for at least one year before randomization for participants <35 years or for at least 6 months for participants ≥35 years (not applicable in case of tubal or severe male factor infertility).
* The trial cycle will be the participant's first controlled ovarian stimulation cycle for IVF/ICSI.
* Regular menstrual cycles of 24-35 days (both inclusive), presumed to be ovulatory.
* Hysterosalpingography, hysteroscopy, saline infusion sonography, or transvaginal ultrasound documenting a uterus consistent with expected normal function (e.g. no evidence of clinically interfering uterine fibroids defined as submucous or intramural fibroids larger than 3 cm in diameter, no polyps and no congenital structural abnormalities which are associated with a reduced chance of pregnancy) within 1 year prior to randomization.
* Transvaginal ultrasound documenting presence and adequate visualisation of both ovaries, without evidence of significant abnormality (e.g. enlarged ovaries which would contraindicate the use of gonadotropins) and normal adnexa (e.g. no hydrosalpinx) within 1 year prior to randomization. Both ovaries must be accessible for oocyte retrieval.
* Early follicular phase (cycle day 2-4) serum levels of FSH between 1 and 15 IU/L (results obtained within 3 months prior to randomization).
* Negative serum Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) antibody tests within 2 years prior to randomization.
* Body mass index (BMI) between 17.5 and 32.0 kg/m2 (both inclusive) at screening.
* Willing to accept transfer of 1-2 embryos.

Exclusion Criteria:

* Known endometriosis stage III-IV (defined by the revised ASRM classification, 1996).
* One or more follicles ≥10 mm (including cysts) observed on the transvaginal ultrasound prior to randomization on stimulation day 1 (puncture of cysts is allowed prior to randomization).
* Known history of recurrent miscarriage (defined as three consecutive losses after ultrasound confirmation of pregnancy (excl. ectopic pregnancy) and before week 24 of pregnancy).
* Known abnormal karyotype of participant or of her partner / sperm donor, as applicable, depending on source of sperm used for insemination in this trial.
* Any known clinically significant systemic disease (e.g. insulin-dependent diabetes).
* Known inherited or acquired thrombophilia disease.
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events.
* Known porphyria.
* Any known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) with the exception of controlled thyroid function disease.
* Known presence of anti-FSH antibodies (based on the information available in the participant's medical records; i.e. not based on the anti-FSH antibody analyses conducted in the trial).
* Known tumours of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus which would contraindicate the use of gonadotropins.
* Known moderate or severe impairment of renal or hepatic function.
* Any abnormal finding of clinical chemistry, haematology or vital signs at screening which is clinically significant as judged by the investigator.
* Currently breast-feeding.
* Undiagnosed vaginal bleeding.
* Known abnormal cervical cytology of clinical significance observed within three years prior to randomization (unless the clinical significance has been resolved).
* Findings at the gynaecological examination at screening which preclude gonadotropin stimulation or are associated with a reduced chance of pregnancy, e.g. congenital uterine abnormalities or retained intrauterine device.
* Pregnancy (negative urinary pregnancy tests must be documented at screening and prior to randomization) or contraindication to pregnancy.
* Known current active pelvic inflammatory disease.
* Use of fertility modifiers during the last menstrual cycle before randomization, including dehydroepiandrosterone (DHEA), metformin or cycle programming with oral contraceptives, progestogen or estrogen preparations.
* Use of hormonal preparations (except for thyroid medication) during the last menstrual cycle before randomization.
* Known history of chemotherapy (except for gestational conditions) or radiotherapy.
* Current or past (1 year prior to randomization) abuse of alcohol or drugs.
* Current (last month) intake of more than 14 units of alcohol per week.
* Current or past (3 months prior to randomization) smoking habit of more than 10 cigarettes per day.
* Hypersensitivity to any active ingredient or excipients in the medicinal products used in the trial.
* Previous participation in the trial.
* Use of any non-registered investigational drugs during the last 3 months prior to randomization.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 1011 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (26):
- China (16):
  - Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing
  - Medical Center for Human Reproduction, Peking University Third Hospital, Beijing
  - Peking University First Hospital, Beijing
  - West China Second University Hospital of Sichuan University, Chengdu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of An'hui Medical University, Hefei
  - Jiangsu Province Hospital, Nanjing
  - ShengJing Hospital of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Tianjin Central Hospital of Gynaecology and Obstetrics, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Renmin Hospital of Wuhan University, Wuhan
  - Tongji Hospital,Tongji Medical College, Huazhong University of Science & Technology, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Vietnam (2):
  - National Center for Assisted Reproductive Technology, Hanoi
  - My Duc Hospital, Ho Chi Minh City

REFERENCES:
- [Result] Qiao J, Zhang Y, Liang X, Ho T, Huang HY, Kim SH, Goethberg M, Mannaerts B, Arce JC. A randomised controlled trial to clinically validate follitropin delta in its individualised dosing regimen for ovarian stimulation in Asian IVF/ICSI patients. Hum Reprod. 2021 Aug 18;36(9):2452-2462. doi: 10.1093/humrep/deab155. PMID 34179971
- [Result] Yang R, Zhang Y, Liang X, Song X, Wei Z, Liu J, Yang Y, Tan J, Zhang Q, Sun Y, Wang W, Qian W, Jin L, Wang S, Xu Y, Yang J, Goethberg M, Mannaerts B, Wu W, Zheng Z, Qiao J. Comparative clinical outcome following individualized follitropin delta dosing in Chinese women undergoing ovarian stimulation for in vitro fertilization /intracytoplasmic sperm injection. Reprod Biol Endocrinol. 2022 Oct 4;20(1):147. doi: 10.1186/s12958-022-01016-y. PMID 36195924
- [Result] Fernandez-Sanchez M, Fatemi H, Garcia-Velasco JA, Heiser PW, Daftary GS, Mannaerts B. Incidence and severity of ovarian hyperstimulation syndrome (OHSS) in high responders after gonadotropin-releasing hormone (GnRH) agonist trigger in "freeze-all" approach. Gynecol Endocrinol. 2023 Dec;39(1):2205952. doi: 10.1080/09513590.2023.2205952. PMID 37156263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 investigational sites randomized participants to the trial: 16 in mainland China, 4 in South Korea, 4 in Taiwan and 2 in Vietnam between Dec 2017 to Jan 2020.
Pre-assignment Details: A total of 1167 participants were screened, wherein, 1011 participants met the eligibility criteria and were randomized. Of these, 1009 participants were exposed to the investigational medicinal product (IMP): 499 participants were exposed to FE 999049 and 510 participants were exposed to GONAL-F. A total of 923 participants completed the trial.
Groups:
- FE 000049 (Follitropin Delta): FE 999049 was administered as single daily subcutaneous injections in the abdomen. Participants randomized to FE 999049 had their individual dose determined on the basis of their anti-Müllerian hormone (AMH) level at screening and their body weight at randomization. The daily FE 999049 dose was fixed throughout the stimulation period and minimum and maximum allowed daily dose was 6 and 12 μg, respectively. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- GONAL-F (Follitropin Alfa): GONAL-F was administered as single daily subcutaneous injections in the abdomen. The starting dose of GONAL-F was 150 IU and fixed for the first five stimulation days, after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 450 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days
Period: Overall Study
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Started (Randomized (2 randomized participants were not exposed to the IMP)) | 500 | 511
Full Analysis Set | 499 | 510
Completed | 465 | 458
Not Completed | 35 | 53
Not completed — Adverse Event | 15 | 33
Not completed — Protocol Deviation | 4 | 0
Not completed — Participant withdrew consent | 3 | 1
Not completed — Discontinuations due to risk of ovarian hyperstimulation syndrome [OHSS] | 9 | 14
Not completed — Discontinuations due to withdrawal from trial | 2 | 3
Not completed — Discontinuations due to thin endometrium or poor endometrial receptivity | 0 | 2
Not completed — Discontinuation due to liquid in uterus | 1 | 0
Not completed — Discontinuation due to risk of Human Immunodeficiency Virus | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) was defined as all randomized and exposed participants. Participants were analyzed according to randomized treatment.
Groups:
- FE 000049 (Follitropin Delta): FE 999049 was administered as single daily subcutaneous injections in the abdomen. Participants randomized to FE 999049 had their individual dose determined on the basis of their AMH level at screening and their body weight at randomization. The daily FE 999049 dose was fixed throughout the stimulation period and minimum and maximum allowed daily dose was 6 and 12 μg, respectively. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- Total: Total of all reporting groups
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa) | Total
Number analyzed (Participants) | 499 | 510 | 1009
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (3.7) | 31.2 (3.8) | 31.1 (3.7)
Age, Customized [Number; unit: years]
  <35 | 394 | 396 | 790
  35-37 | 85 | 86 | 171
  38-40 | 20 | 28 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 499 | 510 | 1009
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 499 | 510 | 1009
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 379 | 381 | 760
  South Korean | 21 | 25 | 46
  Vietnamese | 49 | 51 | 100
  Taiwanese | 50 | 53 | 103
Region of Enrollment [Number; unit: participants]
  China | 378 | 381 | 759
  South Korea | 21 | 25 | 46
  Vietnam | 49 | 51 | 100
  Taiwan | 51 | 53 | 104
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.8 (2.7) | 21.8 (2.8) | 21.8 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy Rate
Description: Defined as at least one intrauterine viable fetus 10-11 weeks after transfer.
Time Frame: 10-11 weeks after transfer
Population: The FAS was defined as all randomized and exposed participants. Participants were analyzed according to randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants | 31.3 | 25.7
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Percentage of participants with ongoing pregnancy rate; Test type: Non-Inferiority — If the lower-limit of the two-sided 95% confidence interval (CI) was greater than the non-inferiority limit (-10.0%), the null hypothesis was rejected. In that case, it would be claimed that FE 999049 was non-inferior to GONAL-F with respect to ongoing pregnancy rate in women undergoing controlled ovarian stimulation; Risk Difference (RD) = 5.4, 95% CI 2-sided [-0.2 to 11.0] — The difference (FE 999049 - GONAL-F) in rates was estimated and a two-sided 95% Cl was constructed using the Mantel-Haenszel method to combine results across age strata

2. Secondary Outcome: Positive Beta Unit of Human Chorionic Gonadotropin (βhCG) Rate
Description: Defined as positive βhCG test 13-15 days after transfer.
Time Frame: 13-15 days after transfer
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants | 41.7 | 35.3
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Percentage of participants with positive beta-hCG; Test type: Other; Risk Difference (RD) = 6.3, 95% CI 2-sided [0.3 to 12.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Clinical Pregnancy Rate
Description: Defined as at least one gestational sac 5-6 weeks after transfer.
Time Frame: 5-6 weeks after transfer
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants | 36.1 | 31.2
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Percentage of participants with at least one gestational sac 5-6 weeks after transfer; Test type: Other; Risk Difference (RD) = 4.9, 95% CI 2-sided [-0.9 to 10.7] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Vital Pregnancy Rate
Description: Defined as at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after transfer.
Time Frame: 5-6 weeks after transfer
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants | 32.3 | 28.0
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Percentage of participants with at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after transfer; Test type: Other; Risk Difference (RD) = 4.2, 95% CI 2-sided [-1.5 to 9.8] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Implantation Rate
Description: Defined as number of gestational sacs 5-6 weeks after transfer divided by number of embryos transferred.
Time Frame: 5-6 weeks after transfer
Population: Participants with embryo transfer (a total of 548 and 546 embryos were transferred in the FE 999049 and GONAL-F groups, respectively). The experimental unit was transferred embryo.
Measure: Number; unit: percentage of sacs/embryos transferred
Units Other Than Participants: Embryos transferred
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
Number analyzed (Embryos transferred) | 548 | 546
percentage of sacs/embryos transferred | 35.6 | 31.3
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Percentage of implanted embryos 5-6 weeks after transfer; Test type: Other; Risk Difference (RD) = 3.9, 95% CI 2-sided [-1.6 to 9.5] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Ongoing Implantation Rate
Description: Defined as number of intrauterine viable fetuses 10-11 weeks after transfer divided by number of embryos transferred.
Time Frame: 10-11 weeks after transfer
Population: Participants with embryo transfer (a total of 548 and 546 embryos were transferred in the FE 999049 and GONAL-F groups, respectively). The experimental unit was transferred embryos.
Measure: Number; unit: % of viable fetus/embryos transferred
Units Other Than Participants: Embryos transferred
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
Number analyzed (Embryos transferred) | 548 | 546
% of viable fetus/embryos transferred | 30.7 | 25.8
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Percentage of participants with ongoing implantation rate; Test type: Other; Risk Difference (RD) = 4.4, 95% CI 2-sided [-0.9 to 9.7] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Proportion of Subjects With Extreme Ovarian Responses
Description: Extreme ovarian response defined as <4, ≥15 or ≥ 20 oocytes retrieved. Participants with cycle cancellation due to poor ovarian response are included as <4 oocytes retrieved.
Time Frame: Oocyte retrieval visit
Population: The FAS was defined as all randomized and exposed participants. Participants analyzed for this endpoint represent participants with oocytes retrieved and participants with cycle cancellation due to poor ovarian response.
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 495 | 507
percentage of participants
  <4 or >=15 oocytes retrieved | 30.3 | 35.1
  <4 or >=20 oocytes retrieved | 17.4 | 18.9
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with <4 or >=15 oocytes retrieved; Test type: Superiority — Logistic regression including AMH group as a factor; p = 0.083, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.60 to 1.03] — Odds ratio is equal to FE 999049/GONAL-F
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with <4 or >=20 oocytes retrieved; Test type: Other — Logistic regression including AMH group as a factor; p = 0.489, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.65 to 1.23] — Odds ratio is equal to FE 999049/GONAL-F

8. Secondary Outcome: Proportion of Subjects With Early OHSS (Including OHSS of Moderate/Severe Grade) and/or Preventive Interventions for Early OHSS
Description: Early OHSS was defined as OHSS with onset ≤9 days after triggering of final follicular maturation. Classification of grade was according to Golan's classification system, and all OHSS cases were graded as mild, moderate or severe.
Time Frame: Up to 9 days after triggering of final follicular maturation
Population: The safety analysis set was defined as all randomized and exposed participants. Participants were analyzed according to actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants
  Early OHSS (any grade) | 4.0 | 6.5
  Early OHSS (moderate/severe) | 3.6 | 4.7
  Any preventive intervention | 1.2 | 3.5
  Early OHSS (any grade) and/or preventive interventions | 5.0 | 9.6
  Early OHSS (moderate/severe) and/or preventive interventions | 4.6 | 7.8
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with early OHSS (any grade); Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p = 0.075, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.34 to 1.06] — Odds ratio is equal to FE 999049/GONAL-F
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with early OHSS (moderate/severe); Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p = 0.365, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.40 to 1.40] — Odds ratio is equal to FE 999049/GONAL-F
Statistical Analysis 3: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with any preventive intervention; Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p = 0.012, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.13 to 0.83] — Odds ratio is equal to FE 999049/GONAL-F
Statistical Analysis 4: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with early OHSS (any grade) and/or preventive interventions; Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p = 0.004, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.30 to 0.81] — Odds ratio is equal to FE 999049/GONAL-F
Statistical Analysis 5: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with early OHSS (moderate/severe) and/or preventive interventions; Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.33 to 0.95] — Odds ratio is equal to FE 999049/GONAL-F

9. Secondary Outcome: Proportion of Subjects With Cycle Cancellation Due to Poor or Excessive Ovarian Response or Embryo Transfer Cancellation Due to Excessive Ovarian Response / OHSS Risk
Description: For each participant the reason for each cycle cancellation was recorded. Embryo transfer cancellation due to adverse events, such as ovarian hyperfunction, OHSS and progesterone increased in participants with embryos available for transfer, were considered as transfer cancellations due to excessive response / OHSS risk.
Time Frame: End-of-stimulation visit (up to 20 days) or transfer visit
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants
  Cycle cancellation due to poor response | 3.4 | 0.8
  Cycle cancellation due to excessive response | 0 | 0
  Transfer cancellation due to excessive ovarian response/ OHSS risk | 5.2 | 12.4
  Cycle cancellation: poor/excessive response, or transfer cancellation excessive response/OHSS risk | 8.6 | 13.1
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with cycle cancellation due to poor response; Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p = 0.002, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 4.58, 95% CI 2-sided [1.52 to 13.74] — Odds ratio is equal to FE 999049/GONAL-F
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with transfer cancellation due to excessive ovarian response/OHSS risk; Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p < 0.001, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.24 to 0.62] — Odds ratio is equal to FE 999049/GONAL-F
Statistical Analysis 3: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Proportion of participants with cycle cancellation due to poor or excessive response, or transfer cancellation due to excessive response/OHSS risk; Test type: Other — Treatment groups were compared using a logistic regression model including age stratum as factor; p = 0.020, Regression, Logistic — The p-value is based on the likelihood ratio test; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.42 to 0.93] — Odds ratio is equal to FE 999049/GONAL-F

10. Secondary Outcome: Number of Follicles on Stimulation Day 6
Description: Counted by ultrasound for the right and left ovary for each participant.
Time Frame: On stimulation Day 6
Population: The FAS was defined as all randomized and exposed participants. Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: number of follicles
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 498 | 509
number of follicles
  Follicles >= 10 mm | 5.4 (3.5) | 6.4 (4.0)
  Follicles >= 12 mm | 2.3 (2.2) | 2.9 (2.5)
  Follicles >= 15 mm | 0.3 (0.7) | 0.3 (0.8)
  Follicles >= 17 mm | 0.1 (0.3) | 0.0 (0.2)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 10 mm; Test type: Superiority; p < .001, van Elteren test — 2-sided; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 12 mm; Test type: Superiority; p < .001, van Elteren test — 2-sided; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 3: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 15 mm; Test type: Superiority; p = 0.568, van Elteren test — 2-sided; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 4: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 17 mm; Test type: Superiority; p = 0.839, van Elteren test — 2-sided; p-value based on van Elteren test adjusted for age stratum

11. Secondary Outcome: Number of Follicles At End-of-stimulation (up to 20 Stimulation Days)
Description: Counted by ultrasound for the right and left ovary for each participant.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: number of follicles
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 494 | 509
number of follicles
  Follicles >= 10 mm | 12.4 (5.6) | 14.2 (6.6)
  Follicles >= 12 mm | 10.3 (4.9) | 11.9 (5.7)
  Follicles >= 15 mm | 6.5 (3.2) | 7.5 (3.5)
  Follicles >= 17 mm | 4.1 (1.8) | 4.5 (2.0)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 10 mm; Test type: Superiority; p < .001, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 12 mm; Test type: Superiority; p < .001, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 3: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 15 mm; Test type: Superiority; p < .001, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 4: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of follicles >= 17 mm; Test type: Superiority; p = 0.011, van Elteren test; p-value based on van Elteren test adjusted for age stratum

12. Secondary Outcome: Size of Follicles on Stimulation Day 6
Description: Counted by ultrasound for the right and left ovary for each participant.
Time Frame: On stimulation Day 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 461 | 493
mm
  Largest follicle (mm) | 13.1 (2.0) | 13.2 (1.8)
  Average follicle size (mm) | 11.5 (1.0) | 11.6 (1.0)
  Average size of 3 largest follicles (mm): number analyzed (Participants) | 393 | 441
  Average size of 3 largest follicles (mm) | 12.5 (1.6) | 12.6 (1.4)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Largest follicle (mm); Test type: Superiority; p = 0.140, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Average follicle size (mm); Test type: Superiority; p = 0.155, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 3: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Treatment comparison: Average size of 3 largest follicles (mm); Test type: Superiority; p = 0.159, van Elteren test; p-value based on van Elteren test adjusted for age stratum

13. Secondary Outcome: Size of Follicles At End-of-stimulation (up to 20 Stimulation Days)
Description: Counted by ultrasound for the right and left ovary for each participant.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 490 | 509
mm
  Largest follicle (mm) | 19.8 (1.9) | 19.8 (1.6)
  Average follicle size (mm) | 15.0 (1.3) | 15.1 (1.1)
  Average size of 3 largest follicles (mm): number analyzed (Participants) | 482 | 505
  Average size of 3 largest follicles (mm) | 18.6 (1.4) | 18.7 (1.1)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Largest follicle (mm); Test type: Superiority; p = 0.848, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Average follicle size (mm); Test type: Superiority; p = 0.629, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 3: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Average size of 3 largest follicles (mm); Test type: Superiority; p = 0.768, van Elteren test; p-value based on van Elteren test adjusted for age stratum

14. Secondary Outcome: Number of Oocytes Retrieved
Description: The number of oocytes retrieved was recorded at the oocyte retrieval visit.
Time Frame: On the day of oocyte retrieval (36 h [±2h] after triggering of final follicular maturation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: oocytes retrieved
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
oocytes retrieved | 10.0 (6.1) | 12.4 (7.3)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Mean number of oocytes retrieved; Test type: Superiority; p < .001, van Elteren test; p-value based on van Elteren test adjusted for age stratum

15. Secondary Outcome: Proportion of Subjects With <4, 4-7, 8-14, 15-19 and ≥20 Oocytes Retrieved
Description: Grouped according to the number of oocytes retrieved. Participants with cycle cancellation due to poor ovarian response are included in the <4 oocytes group.
Time Frame: On the day of oocyte retrieval
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 495 | 507
percentage of participants
  <4 (low response) | 11.3 | 4.7
  4 -7 (moderate response) | 23.0 | 22.3
  8-14 (targeted response) | 46.7 | 42.6
  15-19(hyperresponse) | 12.9 | 16.2
  >=20 (severe hyperresponse) | 6.1 | 14.2

16. Secondary Outcome: Percentage of Metaphase II (MII) Oocytes
Description: The percentage of MII oocytes to oocytes retrieved for participants where all oocytes were inseminated using intracytoplasmic sperm injection (ICSI) are presented.
Time Frame: Prior to insemination
Population: The FAS was defined as all randomized and exposed participants. Participants analyzed for this endpoint represent participants with all oocytes inseminated using ICSI.
Measure: Mean (Standard Deviation); unit: percentage of oocytes
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 223 | 232
percentage of oocytes | 79.5 (17.6) | 77.8 (17.7)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Percentage of MII oocytes / oocytes retrieved; Test type: Superiority; p = 0.197, van Elteren test; p-value based on van Elteren test adjusted for age stratum

17. Secondary Outcome: Fertilization Rate
Description: The fertilization rate was defined as the number of oocytes with 2 pronuclei divided by the number of oocytes retrieved.
Time Frame: On Day 1 after oocyte retrieval
Population: Participants with oocytes retrieved.
Measure: Mean (Standard Deviation); unit: percentage of fertilized oocytes
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 477 | 502
percentage of fertilized oocytes | 63.5 (22.9) | 63.9 (21.0)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Fertilization rate relative to oocytes retrieved; Test type: Superiority; p = 0.790, van Elteren test; p-value based on van Elteren test adjusted for age stratum

18. Secondary Outcome: Number and Quality of Embryos
Description: Number of embryos (total and good-quality) on Day 3 are presented. A good-quality embryo was defined as an embryo with ≥6 blastomeres and ≤20% fragmentation, without signs of multinucleation.
Time Frame: On Day 3 after oocyte retrieval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
embryos
  Number of embryos | 7.0 (4.6) | 8.7 (5.5)
  Number of good-quality embryos | 4.1 (3.6) | 5.2 (4.3)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of embryos on day 3; Test type: Superiority; p < .001, van Elteren test; p-value based on van Elteren test adjusted for age stratum
Statistical Analysis 2: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of good-quality embryos on Day 3; Test type: Superiority; p < .001, van Elteren test; p-value based on van Elteren test adjusted for age stratum

19. Secondary Outcome: Circulating Concentrations of Luteinizing Hormone (LH)
Description: Blood samples for analysis of circulating concentrations of LH were drawn. The median and inter-quartile range (IQR) of LH levels on stimulation Day 6 are presented.
Time Frame: On stimulation Day 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 496 | 508
IU/L | 2.6 [1.7 to 4.7] | 3.1 [1.9 to 6.8]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of LH on stimulation Day 6; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.81, 95% CI 2-sided [0.74 to 0.88] — Mean ratio is equal to FE 999049/GONAL-F

20. Secondary Outcome: Circulating Concentrations of LH
Description: Blood samples for analysis of circulating concentrations of LH were drawn. The median and IQR of LH levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 492 | 503
IU/L | 1.8 [1.1 to 2.9] | 2.0 [1.2 to 3.1]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of LH at end-of-stimulation; Test type: Superiority; p = 0.018, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.90, 95% CI 2-sided [0.82 to 0.98]

21. Secondary Outcome: Circulating Concentrations of Estradiol
Description: Blood samples for analysis of circulating concentrations of estradiol were drawn. The median and IQR of estradiol levels on stimulation Day 6 are presented.
Time Frame: On stimulation Day 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 497 | 509
pmol/L | 2240.7 [1325.8 to 3641.1] | 2885.9 [1729.4 to 4492.1]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Estradiol on stimulation Day 6; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.77, 95% CI 2-sided [0.70 to 0.84] — Mean ratio is equal to FE 999049/GONAL-F

22. Secondary Outcome: Circulating Concentrations of Estradiol
Description: Blood samples for analysis of circulating concentrations of estradiol were drawn. The median and IQR of estradiol levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 491 | 504
pmol/L | 7429.3 [4786.2 to 10439.8] | 9055.8 [6214.2 to 12964.3]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Estradiol at end-of-stimulation; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.74, 95% CI 2-sided [0.68 to 0.81] — Mean ratio is equal to FE 999049/GONAL-F

23. Secondary Outcome: Circulating Concentrations of Progesterone
Description: Blood samples for analysis of circulating concentrations of progesterone were drawn. The median and IQR of progesterone levels on stimulation Day 6 are presented.
Time Frame: On stimulation Day 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 497 | 507
nmol/L | 1.7 [0.8 to 2.6] | 1.9 [0.8 to 2.9]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Progesterone on stimulation Day 6; Test type: Superiority; p = 0.003, ANCOVA — The p-value corresponds to the two-sided F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean Ratio = 0.89, 95% CI 2-sided [0.82 to 0.96] — Mean ratio is equal to FE 999049/GONAL-F

24. Secondary Outcome: Circulating Concentrations of Progesterone
Description: Blood samples for analysis of circulating concentrations of progesterone were drawn. The median and IQR of progesterone levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 490 | 502
nmol/L | 2.4 [1.7 to 3.5] | 3.2 [2.2 to 4.4]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Progesterone at end-of-stimulation; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.74, 95% CI 2-sided [0.68 to 0.79] — Mean ratio is equal to FE 999049/GONAL-F

25. Secondary Outcome: Circulating Concentrations of Inhibin A
Description: Blood samples for analysis of circulating concentrations of inhibin A. The median and IQR of inhibin A levels on stimulation Day 6 are presented.
Time Frame: On stimulation Day 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 496 | 508
ng/L | 107.9 [61.6 to 163.5] | 129.1 [84.6 to 203.6]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Inhibin A on stimulation Day 6; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.76, 95% CI 2-sided [0.70 to 0.83]

26. Secondary Outcome: Circulating Concentrations of Inhibin A
Description: Blood samples for analysis of circulating concentrations of inhibin A were drawn. The median and IQR of inhibin A levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 491 | 504
ng/L | 361.7 [252.8 to 525.6] | 447.4 [307.5 to 630.9]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Inhibin A at end-of-stimulation; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.77, 95% CI 2-sided [0.71 to 0.83] — Mean ratio is equal to FE 999049/GONAL-F

27. Secondary Outcome: Circulating Concentrations of Inhibin B
Description: Blood samples for analysis of circulating concentrations of Inhibin B were drawn. The median and IQR of inhibin B levels on stimulation Day 6 are presented.
Time Frame: On stimulation Day 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 445 | 452
ng/L | 740.0 [481.0 to 1069.0] | 901.0 [588.0 to 1317.5]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Inhibin B on stimulation Day 6; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.83, 95% CI 2-sided [0.77 to 0.89] — Mean ratio is equal to FE 999049/GONAL-F

28. Secondary Outcome: Circulating Concentrations of Inhibin B
Description: Blood samples for analysis of circulating concentrations of Inhibin B were drawn. The median and IQR of inhibin B levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 445 | 449
ng/L | 1020.0 [689.0 to 1488.0] | 1101.0 [738.0 to 1665.0]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of Inhibin B at end-of-stimulation; Test type: Superiority; p = 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.87, 95% CI 2-sided [0.80 to 0.95] — Mean ratio is equal to FE 999049/GONAL-F

29. Secondary Outcome: Circulating Concentrations of Follicle-stimulating Hormone (FSH)
Description: Blood samples for analysis of circulating concentrations of FSH were drawn. The median and IQR of FSH levels on stimulation Day 6 are presented.
Time Frame: On stimulation Day 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 497 | 509
IU/L | 11.6 [9.5 to 14.8] | 11.2 [9.5 to 13.3]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of FSH on stimulation Day 6; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 1.08, 95% CI 2-sided [1.04 to 1.12] — Mean ratio is equal to FE 999049/GONAL-F

30. Secondary Outcome: Circulating Concentrations of FSH
Description: Blood samples for analysis of circulating concentrations of FSH were drawn. The median and IQR of FSH levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 491 | 504
IU/L | 11.3 [9.2 to 14.4] | 12.2 [10.4 to 15.2]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of FSH at end-of-stimulation; Test type: Superiority; p < 0.001, ANCOVA — The p-value corresponds to F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 0.92, 95% CI 2-sided [0.89 to 0.95] — Mean ratio is equal to FE 999049/GONAL-F

31. Secondary Outcome: Circulating Concentrations of FSH
Description: Blood samples for analysis of circulating concentrations of FSH were drawn. The median and IQR of FSH levels at oocyte retrieval are presented.
Time Frame: At oocyte retrieval
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 478 | 503
IU/L | 5.6 [4.5 to 7.1] | 5.5 [4.4 to 6.9]
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Circulating concentrations of FSH at oocyte retrieval visit; Test type: Superiority; p = 0.184, ANCOVA — The p-value corresponds to the two-sided F-test of treatment effect; The multiplicative ANCOVA model included treatment and age stratum as fixed factors; Mean ratio = 1.03, 95% CI 2-sided [0.99 to 1.07] — Mean ratio is equal to FE 999049/GONAL-F

32. Secondary Outcome: Total Gonadotropin Dose
Description: Calculated by start dates, end dates and daily dose of IMP.
Time Frame: Up to 20 stimulation days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram of dose
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
microgram of dose | 77.5 (24.4) | 109.9 (32.9)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Total gonadotropin dose; Test type: Superiority; p < .001, van Elteren test; p-value is based on van Elteren test adjusted for AMH group

33. Secondary Outcome: Proportion of Subjects With Investigator-requested Gonadotropin Dose Adjustments
Description: Investigator-requested decreases and increases of the gonadotropin dose were captured during the stimulation period.
Time Frame: Up to 20 stimulation days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants | 57.1 | 55.3

34. Secondary Outcome: Number of Stimulation Days
Description: Calculated by start dates and end dates.
Time Frame: Up to 20 stimulation days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
days | 9.2 (1.9) | 8.7 (1.6)
Statistical Analysis 1: Comparison: FE 000049 (Follitropin Delta) vs GONAL-F (Follitropin Alfa); Number of stimulation days; Test type: Superiority — Treatment groups were compared using the van Elteren test; p = 0.001, van Elteren; p-value is based on van Elteren test adjusted for AMH group

35. Secondary Outcome: Number of Participants With Adverse Events
Description: Any adverse event occurring after start of IMP and before the end-of-trial visit, or a pre-treatment adverse event or pre-existing medical condition that worsens in intensity after start of IMP and before the end-of-trial visit was considered treatment-emergent, and is presented for this endpoint.
Time Frame: From screening up to end-of-trial (up to approximately 5.5 months)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 449 | 510
percentage of participants | 46.3 | 43.1

36. Secondary Outcome: Intensity of Adverse Events
Description: The intensity of adverse event was classified using the following 3-point scale: mild = awareness of signs or symptoms, but no disruption of usual activity; moderate = event sufficient to affect usual activity (disturbing); or severe = inability to work or perform usual activities (unacceptable).
Time Frame: From screening up to end-of-trial (up to approximately 5.5 months)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants
  Mild adverse events | 40.1 | 37.8
  Moderate adverse events | 7.4 | 5.9
  Severe adverse events | 3.6 | 1.8

37. Secondary Outcome: Changes From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase and Gamma Glutamyl Transferase
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Alanine aminotransferase, Alkaline phosphatase, Aspartate aminotransferase and Gamma glutamyl transferase.
Time Frame: From screening up to end-of-trial (up to approximately 5.5 months)
Population: The safety analysis set was defined as all randomized and exposed participants. Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 494 | 506
IU/L
  Alanine aminotransferase: number analyzed (Participants) | 493 | 501
  Alanine aminotransferase | 3.9 (13.8) | 4.6 (16.7)
  Alkaline phosphatase | -2.9 (8.2) | -2.7 (8.0)
  Aspartate aminotransferase: number analyzed (Participants) | 490 | 496
  Aspartate aminotransferase | 0.7 (7.1) | 1.2 (13.0)
  Gamma glutamyl transferase | 1.1 (6.6) | 1.1 (10.2)

38. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Bicarbonate, Blood Urea Nitrogen, Calcium, Chloride, Cholesterol, Glucose, Phosphate, Potassium and Sodium
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Bicarbonate, Blood urea nitrogen, Calcium, Chloride, Cholesterol, Glucose, Phosphate, Potassium and Sodium.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 494 | 506
mmol/L
  Bicarbonate: number analyzed (Participants) | 493 | 503
  Bicarbonate | -0.83 (2.52) | -0.72 (2.51)
  Blood urea nitrogen | -0.27 (1.12) | -0.23 (1.11)
  Calcium | -0.010 (0.089) | 0.000 (0.081)
  Chloride | -0.3 (2.3) | -0.3 (2.4)
  Cholesterol | 0.218 (0.537) | 0.260 (0.549)
  Glucose: number analyzed (Participants) | 493 | 503
  Glucose | -0.01 (0.94) | -0.01 (0.91)
  Phosphate | 0.037 (0.166) | 0.023 (0.169)
  Potassium: number analyzed (Participants) | 494 | 504
  Potassium | 0.03 (0.34) | 0.04 (0.33)
  Sodium | -1.8 (2.6) | -1.7 (2.5)

39. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Albumin and Protein.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 494 | 506
g/L
  Albumin | -2.0 (3.1) | -1.6 (3.0)
  Protein | -2.3 (4.6) | -1.5 (4.5)

40. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Lactate Dehydrogenase
Description: Blood samples were collected for the analysis of clinical chemistry parameter including: Lactate dehydrogenase.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 452 | 455
U/L | -3.0 (17.0) | -0.9 (18.9)

41. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Direct Bilirubin, Bilirubin, Creatinine, Urate
Description: Blood samples were collected for the analysis of clinical chemistry parameter including: Direct bilirubin, Bilirubin, Creatinine, Urate.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 494 | 506
umol/L
  Direct bilirubin: number analyzed (Participants) | 478 | 480
  Direct bilirubin | -0.3 (0.8) | -0.2 (0.8)
  Bilirubin: number analyzed (Participants) | 493 | 503
  Bilirubin | -1.3 (3.6) | -1.0 (3.5)
  Creatinine | -3.4 (9.0) | -3.5 (8.5)
  Urate | -18.8 (54.1) | -17.9 (53.5)

42. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes of Clinical Chemistry: Alanine Aminotransferase, Aspartate Aminotransferase, Bicarbonate, Calcium, Phosphate
Description: The table represents the percentage of participants in each group with normal baseline values and markedly abnormal end-of-stimulation or end-of-trial values for alanine aminotransferase, aspartate aminotransferase, bicarbonate, calcium, phosphate.
Time Frame: End-of-stimulation visit and end-of-trial visit
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 494 | 505
percentage of participants
  Alanine aminotransferase (IU/L) (End-of-stimulation): number analyzed (Participants) | 484 | 477
  Alanine aminotransferase (IU/L) (End-of-stimulation) | 0.2 | 0.2
  Aspartate aminotransferase (IU/L) (End-of-stimulation): number analyzed (Participants) | 484 | 484
  Aspartate aminotransferase (IU/L) (End-of-stimulation) | 0 | 0.2
  Phosphate (mmol/L) (End-of-stimulation): number analyzed (Participants) | 489 | 501
  Phosphate (mmol/L) (End-of-stimulation) | 0.2 | 0.0
  Alanine aminotransferase (IU/L) (End-of-trial): number analyzed (Participants) | 488 | 480
  Alanine aminotransferase (IU/L) (End-of-trial) | 0.4 | 0.6
  Bicarbonate (mmol/L) (End-of-trial): number analyzed (Participants) | 478 | 492
  Bicarbonate (mmol/L) (End-of-trial) | 1.3 | 0.8
  Calcium (mmol/L) (End-of-trial) | 0 | 0.2

43. Secondary Outcome: Change From Baseline in Haematology Parameter: Erythrocytes
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocytes.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 489 | 503
10^12 cells/L | -0.13 (0.31) | -0.09 (0.27)

44. Secondary Outcome: Change From Baseline in Haematology Parameters: Leukocytes and Platelets
Description: Blood samples were collected for the analysis of haematology parameters including: Leukocytes and Platelets.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 489 | 503
10^9 cells/L
  Leukocytes | 1.161 (2.232) | 0.996 (2.099)
  Platelets: number analyzed (Participants) | 483 | 495
  Platelets | 19.9 (41.7) | 23.8 (40.6)

45. Secondary Outcome: Change From Baseline in Haematology Parameter: Haemoglobin
Description: Blood samples were collected for the analysis of haematology parameter including: Haemoglobin.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 489 | 503
g/L | -2.9 (8.9) | -1.7 (7.9)

46. Secondary Outcome: Change From Baseline in Haematology Parameter: Haematocrit
Description: Blood samples were collected for the analysis of haematology parameter including: Haematocrit.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 480 | 491
Ratio | -0.012 (0.033) | -0.008 (0.030)

47. Secondary Outcome: Change From Baseline in Haematology Parameter: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocyte mean corpuscular volume.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 480 | 491
Femtoliters | 0.0 (3.3) | 0.1 (3.2)

48. Secondary Outcome: Change From Baseline in Haematology Parameter: Erythrocyte Mean Corpuscular Haemoglobin
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocyte mean corpuscular haemoglobin.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 489 | 503
picogram | 0.3 (0.9) | 0.2 (0.8)

49. Secondary Outcome: Change From Baseline in Haematology Parameter: Erythrocyte Mean Corpuscular Haemoglobin Concentration
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocyte mean corpuscular haemoglobin concentration.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 480 | 491
mmol/L | 0.2 (0.8) | 0.1 (0.8)

50. Secondary Outcome: Change From Baseline in Haematology Parameters: Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes and Neutrophils/Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters including: Basophils/leukocytes, Eosinophils/leukocytes, Lymphocytes/leukocytes, Monocytes/leukocytes and Neutrophils/leukocytes.
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 489 | 502
percentage
  Basophils/leukocytes | -0.01 (0.37) | 0.02 (0.36)
  Eosinophils/leukocytes | -0.01 (1.08) | -0.07 (1.04)
  Lymphocytes/leukocytes | -2.05 (9.18) | -1.39 (9.16)
  Monocytes/leukocytes | -0.16 (1.52) | -0.04 (1.66)
  Neutrophils/leukocytes | 2.20 (10.03) | 1.50 (9.89)

51. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes of Haematology Parameters: Leukocytes, Lymphocytes/Leukocytes
Description: The table represents the percentage of participants in each group with normal baseline values and markedly abnormal end-of-stimulation and end-of-trial values for leukocytes and lymphocytes/leukocytes.
Time Frame: End-of-stimulation visit and end-of-trial visit
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 474 | 487
percentage of participants
  Leukocytes (10^9 cells/L) (End-of-stimulation): number analyzed (Participants) | 455 | 460
  Leukocytes (10^9 cells/L) (End-of-stimulation) | 0.7 | 0
  Lymphocytes/leukocytes (%) (End-of-stimulation): number analyzed (Participants) | 471 | 481
  Lymphocytes/leukocytes (%) (End-of-stimulation) | 0.4 | 0.2
  Leukocytes (10^9 cells/L) (End-of-trial): number analyzed (Participants) | 459 | 468
  Leukocytes (10^9 cells/L) (End-of-trial) | 0.7 | 0
  Lymphocytes/leukocytes (%) (End-of-trial) | 0.6 | 0

52. Secondary Outcome: Number of Immune-related Adverse Events
Description: Standardised Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQs).
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 8
Measure: Number; unit: events
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
events | 0 | 0

53. Secondary Outcome: Frequency of Injection Site Reactions
Description: Assessed by the participant during the stimulation period. Participants assessed the injection site reactions (redness, pain, itching, swelling and bruising) three times daily: immediately after the injection, 30 minutes after the injection and 24 hours after the injection.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants | 23.2 | 21.6

54. Secondary Outcome: Intensity of Injection Site Reactions
Description: Assessed by the participant during the stimulation period as mild, moderate or severe. Participants are tabulated according to the highest severity of their reported injection site reactions.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants
  Mild injection site reaction | 21.6 | 21.2
  Moderate injection site reaction | 1.6 | 0.4
  Severe injection site reaction | 0 | 0

55. Secondary Outcome: Proportion of Subjects With Treatment-induced Anti-FSH Antibodies, Overall as Well as With Neutralizing Capacity
Description: Measured by presence of anti-FSH antibodies.
Time Frame: Up to 28 days after end of the stimulation period
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants
  Treatment-induced anti-FSH antibodies (Overall) | 1.40 [0.57 to 2.87] | 0.98 [0.32 to 2.27]
  Treatment-induced anti-FSH antibodies with neutralizing capacity | 0 [NA to NA] — For participants with treatment-induced anti-FSH antibodies, none of the antibodies were of neutralizing capacity at any sampling time point. | 0 [NA to NA] — For participants with treatment-induced anti-FSH antibodies, none of the antibodies were of neutralizing capacity at any sampling time point.

56. Secondary Outcome: Intensity of Immune-related Adverse Events
Description: The intensity of immune-related adverse event was classified using the following 3-point scale: mild = awareness of signs or symptoms, but no disruption of usual activity; moderate = event sufficient to affect usual activity (disturbing); or severe = inability to work or perform usual activities (unacceptable).
Time Frame: From screening up to end-of-trial (approximately 5.5 months)
Population: as for outcome 8
Measure: Number; unit: events
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
events
  Mild | 0 | 0
  Moderate | 0 | 0
  Severe | 0 | 0

57. Secondary Outcome: Proportion of Subjects With Cycle Cancellations Due to an Adverse Event, Including Immune-related Adverse Events, or Due to Technical Malfunctions of the Administration Pen
Description: For each participant the reason for cycle cancellation will be recorded.
Time Frame: Up to 20 stimulation days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants
  Adverse event (including immune-related adverse events) | 0 | 0.2
  Technical malfunctions of the administration pen | 0 | 0

58. Secondary Outcome: Proportion of Subjects With Late OHSS
Description: Late OHSS was defined as OHSS with onset >9 days after triggering of final follicular maturation. The proportion of participants with late OHSS, and late OHSS of moderate or severe grade are presented. All OHSS cases were graded as mild, moderate, or severe.
Time Frame: After 9 days post triggering of final follicular maturation
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants
  Late OHSS (Any grade) | 4.0 | 2.0
  Late OHSS (Moderate/severe) | 3.6 | 1.8

59. Secondary Outcome: Proportion of Participants With Multi-fetal Gestation
Description: Defined as pregnancy with more than one fetus. Among participants with ongoing pregnancy, percentage of participants with twin pregnancies are presented.
Time Frame: End-of-trial
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 156 | 131
percentage of participants | 7.7 | 9.9

60. Secondary Outcome: Proportion of Participants With Early Pregnancy Losses
Description: Grouped according to occurrence of biochemical pregnancy, spontaneous abortion, vanishing twin or ectopic pregnancy (with and without medical/surgical intervention).
  Frequency of early pregnancy losses are presented.
Time Frame: End-of-trial
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 208 | 180
percentage of participants | 25.0 | 27.2

61. Secondary Outcome: Proportion of Participants With Technical Malfunctions of the Administration Pen
Description: Incidences of technical malfunctions of the administration pen were recorded.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 499 | 510
percentage of participants | 0.4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from screening up to end-of-trial (up to approximately 5.5 months).
Description: Any adverse event occurring after start of IMP and before the end-of-trial visit, or a pre-treatment adverse event or pre-existing medical condition that worsens in intensity after start of IMP and before the end-of-trial visit were considered treatment-emergent and are presented for the safety analysis set.
  The safety analysis set was defined as all randomized and exposed participants. Participants were analyzed according to actual treatment received.
Arm/Group | FE 000049 (Follitropin Delta) | GONAL-F (Follitropin Alfa)
All-Cause Mortality (participants affected / at risk) | 0/499 | 0/510
Serious Adverse Events (participants affected / at risk) | 30/499 | 18/510
Other Adverse Events (participants affected / at risk) | 97/499 | 94/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 000049 (Follitropin Delta) (N=499) | GONAL-F (Follitropin Alfa) (N=510)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 11 (11) | 8 (8)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 000049 (Follitropin Delta) (N=499) | GONAL-F (Follitropin Alfa) (N=510)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 29 (29) | 35 (35)
Pelvic discomfort (Reproductive system and breast disorders) | 25 (26) | 28 (30)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 25 (25) | 21 (21)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 25 (25) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (3):
  • Study Protocol: Protocol excluding mainland China (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03296527/Prot_000.pdf
  • Study Protocol: Protocol specific for mainland China (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03296527/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT03296527/SAP_002.pdf